CLINICAL TRIAL: NCT02739386
Title: Evaluation of Hospitalization for Complications of Autoimmune Disease Following Ipilimumab Treatment Among Melanoma Patients With Underlying Autoimmune Diseases Treated in Routine Clinical Practices in the US
Brief Title: Study of Autoimmune Disease Complications Following Ipilimumab Treatment Among Melanoma Patients With Underlying Autoimmune Diseases
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA184-486
Record Dates: First submitted 2016-04-07; First posted 2016-04-15 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort Population: Individuals included in a large US-based administrative medical claims database with underlying autoimmune disorder exposed to ipilimumab for the treatment of melanoma.
  Interventions: Biological: Ipilimumab

INTERVENTIONS:
Biological: Ipilimumab — Intravenous monoclonal antibody injection
  Other Names: Yervoy®

SUMMARY:
The research questions to be addressed by this study are as follows:

1. What is the prevalence of ipilimumab use among adults with a history of autoimmune disease that received treatment with ipilimumab for advanced melanoma?
2. Do melanoma patients with a history of autoimmune disease experience complications that require hospitalization related to their underlying autoimmune disease following treatment with ipilimumab?

ELIGIBILITY:
Inclusion Criteria:

* Received ipilimumab therapy between 03/01/2011 and 6/30/2014
* Aged 18 years or older at index date (initiation of ipilimumab)
* Diagnosed with melanoma before index
* Documented history of an autoimmune disease
* Have at least 6 months of continuous pharmaceutical and medical benefit enrollment prior to the index
* Have at least 3 months of continuous pharmaceutical and medical benefit enrollment following and including the index date

Exclusion Criteria:

* Diagnosed with melanoma but NO record of exposure to ipilimumab
* No exposure to nivolumab (Opdivo ®) at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with an underlying autoimmune disease treated with ipilimumab for advanced melanoma.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Incidence of ipilimumab treatment among adult melanoma patients with a prior or existing autoimmune disease/condition | Approximately 40 months
Incidence of hospitalizations related to the pre-existing autoimmune disease/condition following treatment with ipilimumab | Approximately 40 months

SECONDARY OUTCOMES:
Incidence rate of hospitalization related to a complication of the underlying autoimmune condition before exposure to ipilimumab treatment | Approximately 40 months
Incidence rate of hospitalization related to a complication of the underlying autoimmune condition after exposure to ipilimumab treatment | Approximately 40 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol-Myers Squibb, Princeton, New Jersey, United States

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx